CLINICAL TRIAL: NCT04460040
Title: Exercise-Induced Metabolic Compensation; a Physiological Adaptive Response to Exercise Training
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Gepner Yftach, Principal investigator, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Metabolism
Record Dates: First submitted 2020-06-29; First posted 2020-07-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Exercise Training
Keywords: Metabolic adaptation; Energy expenditure; Exercise; Muscle
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 16 overweight (body mass index: 25-30 kg/m2) men (n=8) and women (n=8) aged 21 to 45 years will exercise for 3 months in a moderate intensity regimen of 20 kcal/week/kg body weight
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Exercise in moderate intensity tailored individually to 20 kcal/kg/week (range 1500-2000 kcal/week) with a free choice to exercise at home/gym on a treadmill or outdoors.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — The first phase of the study will comprise two weeks of control phase when participants will not engage in any exercise training but will be monitored for total daily energy expenditure and its components (REE, SMR, and DIT) and assessed volume of metabolic organs and skeletal muscle efficiency.
  Next, participants will start the active phase. In the first two weeks, participants will perform 150 - 200 min/week of a moderate intensity exercise so that they can adapt to the new regime and avoid injury. All exercise training will be monitored using heart rate sensor (HR) to track exercise adherence and HR range goals. Changes in daily non-exercise physical activity and sedentary behavior will be assessed for 10 days pre- and post-intervention by a tri-axial accelerometer. All study participants will be instructed to consume their habitual diet and to maintain the same caloric intake.

SUMMARY:
The primary aim of this proposal is to identify changes in the volume of highly metabolic organs (liver, kidneys, and brain) that occur as a physiological adaptation to exercise training and lower the resting energy expenditure. Secondary aims are to identify changes in the metabolic efficiency of muscle in low levels of physical activity and evaluate the effects on components of total daily energy expenditure including the sleeping metabolic rate (SMR) and diet induced thermogenesis (DIT).

DETAILED DESCRIPTION:
Using a clinical trial type protocol, 16 overweight (body mass index: 25-30 kg/m2) men (n=8) and women (n=8) aged 21 to 45 years will exercise for 3 months in a moderate intensity regimen of 20 kcal/week/kg body weight that reflects current recommendations for weight management. The volume of various organs will be measured pre- and post-exercise intervention using magnetic resonance imaging (MRI). A cycling ergometer with a varied workload will be used to assess muscle metabolic efficiency. Changes in overnight SMR and 4 hours post breakfast DIT will be evaluated by whole human room indirect calorimetry ("metabolic chamber"). In addition, free-living Total Energy Expenditure (TEE) will be measured for ten days pre- and post-intervention by doubly labeled water.

ELIGIBILITY:
Inclusion Criteria:

Overweight [body mass index (BMI) 25-30

Exclusion Criteria:

* Participation in another exercise or weight loss program in the last 6 months
* Non-stable weight (>±5%) over the past 6 months
* Current regular exercise > 1 hour per week
* Smoking within the past 6 months
* Being post-menopausal, breastfeeding, pregnancy, or having been pregnant within the past 6 months
* Previous bariatric surgery
* Cardiopulmonary disease (e.g., recent myocardial infarction or unstable angina)
* Musculoskeletal or neuromuscular impairments that preclude exercise training
* Having other health issues include cancer, diabetes, thyroid disease, hypertension, chronic renal failure, cognitive impairments
* Use of drugs that potentially impact body metabolism.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-03-27 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
To examine long-term changes in the volume of highly metabolic organs (brain, liver, and kidneys) as an adaptive metabolic response to exercise training | Pre- and post 12 weeks of exercise intervention
  The volume of various organs will be measured using magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
To evaluate the changes in skeletal muscle metabolic efficiency during non- exercise physical activity as an adaptive response to long-term exercise training | Pre- and post 12 weeks of exercise intervention
  A cycling ergometer with a varied workload will be used to assess muscle metabolic efficiency
To determine the effect of long-term exercise training on changes in sleeping metabolic rate as an adaptive response . | Pre- and post 12 weeks of exercise intervention
  Changes in overnight sleeping metabolic rate will be evaluated by whole human room indirect calorimetry ("metabolic chamber")
To assess the effect of long-term exercise training on changes in diet induced thermogenesis as an adaptive response. | Pre- and post 12 weeks of exercise intervention
  Changes in diet induced thermogenesis will be evaluated 4 hours post breakfast by whole human room indirect calorimetry ("metabolic chamber")

CONTACTS AND LOCATIONS:
Overall Officials: Yftach Gepner, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Other, Israel